CLINICAL TRIAL: NCT02763163
Title: Examination of the Link Between Sun Exposure Routine and Bacteria Population of the Skin
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute for Skin Research, Israel (Industry)
Collaborators: Fischer Pharmaceuticals Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1059/15
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- outdoor workers: Subjects with an excessive exposure to the sun on a daily basis
  Interventions: Behavioral: Sun exposure routine
- office workers: Subjects who spend most of the day in a closed shaded room
  Interventions: Behavioral: Sun exposure routine

INTERVENTIONS:
Behavioral: Sun exposure routine

SUMMARY:
These days many studies are conducted testing the symbiosis between the bacteria population to the human body's functioning. The research of the connection between the skin condition and the bacteria population is in its early stages. There is a characterization of different bacteria for different body areas depending on their composition, humidity etc. In addition, there are preliminary findings of biological receptors that react to the contact with bacteria on the surface of the skin and turn on the immune system, awakening it to cope with the new invader. Based on the above information, the investigators hypothesis is that there is a connection between the degrees of sun exposure of individuals to the growing of beneficial bacteria populations on the surface of the skin. The study will compare between the bacteria population on the skin of Israeli subjects, divided to two groups, one with an excessive exposure to the sun on a daily basis, (such as agricultural workers, lifeguards, construction, etc.), and the other of the office worker who spend most of the day in a closed shaded room.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the age of 20-60.

Exclusion Criteria:

* Pregnant or lactating women.
* Volunteers with a known allergy to one of the tested materials or to their ingredients.
* Treatment with medication such as anti-inflammatories, antihistamines,corticosteroids, systemically or topically applied, unless stopped for 2 weeks prior to the trial in the case of systemic treatment and 3 days in the case of topical treatment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Scanning the bacteria population of the surface of the skin by using swab on the cheek area. The samples of bacteria will be characterized by genetic sequencing. | 6 months

IPD SHARING:
Plan to Share IPD: No